CLINICAL TRIAL: NCT03247023
Title: Long Term Follow-up of Integra® Cadence™ Total Ankle System in Primary Ankle Joint Replacement
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision not related to safety
Sponsor: Smith & Nephew, Inc. (Industry)
Collaborators: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Other Study IDs: T-CTAS-002
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-12

CONDITIONS: Degenerative Arthritis; Rheumatoid Arthritis; Traumatic Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Integra Cadence Total Ankle System
  Interventions: Device: Implantation of Integra Cadence Total Ankle Sysyem

INTERVENTIONS:
Device: Implantation of Integra Cadence Total Ankle Sysyem — Primary Ankle Arthroplasty

SUMMARY:
This study will evaluate the long term performance and safety data for the Cadence™ Total Ankle System (CTAS) when used for primary arthroplasty in patients with primary arthritis (e.g. degenerative disease), secondary arthritis (e.g. post-traumatic, avascular necrosis, if minimally 2/3 of the talus is preserved), and systemic arthritis of the ankle (e.g. rheumatoid arthritis, hemochromatosis)

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included if he/she:

* Qualifies for primary Total Ankle Replacement (TAR) per the surgeon and has a diagnosis of one of the following: primary arthritis (e.g. degenerative disease), secondary arthritis (e.g. post-traumatic, avascular necrosis, if minimally 2/3 of the talus is preserved), or systemic arthritis of the ankle (e.g. rheumatoid arthritis, hemochromatosis).
* Is suitable for TAR with Cadence™ Total Ankle System per the study surgeon based on the product indication and having considered deformity, stability, bone quality, soft- tissue envelope, and neurovascular status.
* Is willing and able to complete scheduled follow-up visits, evaluations and questionnaires as described in the Informed Consent (or Information Letter and Data Transfer Authorization Form, as applicable).

Exclusion Criteria:

Subjects will be excluded from the study if he/she:

* Is morbidly obese (defined by a Body Mass Index (BMI) > 40 or BMI of 35 - 40 with significant medical problems caused by or made worse by their weight).
* Has one of the following conditions, which could compromise the affected limb: ankle arthrodesis with malleolar exeresis, severe neurological (Charcot's Arthropathy) or vascular disease, loss of musculature or neuromuscular compromise.
* Has an active local/systemic infection that may affect the prosthetic joint or has a recent history of infection.
* Has a condition that may impair proper wound healing (e.g., poor soft tissue envelope).
* Has a metabolic disorder or disease that may compromise bone quality (e.g. arthrogryposis etc.), physiological or anatomical anomalies, and/or malignancy/local bone tumors.
* Has inadequate neuromuscular status (e.g., prior paralysis, severe neuropathy).
* Has a known sensitivity or allergic reaction to one or more of the implanted materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with ankle arthritis requiring total ankle replacement
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Implant survivorship | 2 years
  Implant survival defined as absence of device removal or revision

SECONDARY OUTCOMES:
Relative change of Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function (PF) - Mobility compared to baseline | up to 10 years
  Relative change of PROMIS PF - Mobility compared to baseline
Relative change of Range of Motion (ROM) compared to baseline | up to 10 years
  Relative change of ROM compared to baseline
Relative change of Foot and Ankle Ability Measure (FAAM) Activities of Daily Living (ADL) subscale compared to baseline | up to 10 years
  Relative change of FAAM ADL compared to baseline
Relative change of Visual Analogue Scale (VAS) Pain compared to baseline | up to 10 years
  Relative change of VAS Pain compared to baseline
Relative change of Quality of Life Measure Short Form - 36v2 (SF-36v2) compared to baseline | up to 10 years
  Relative change of SF-36v2 compared to baseline
Implant survivorship | 5 and 10 years
  Implant survival defined as absence of device removal or revision
Radiographic Success | up to 10 years
  Radiographic success as defined as absence of implant radiolucency, subsidence, tilting, migration defined as no evidence of radiolucency >4 mm in more than 3 zones and of subsidence or tilting ˃4 degrees, or migration > 4mm

CONTACTS AND LOCATIONS:
Locations (6):
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - Foot and Ankle Institute, Woluwe-St-Lambert
- St. Michael's Hospital, Toronto, Canada
- CHRU Tours, Tours, France
- Clinica Nostra Senhora del Remei, Barcelona, Spain
- North Cumbria University Hospitals, Carlisle, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided